CLINICAL TRIAL: NCT03288558
Title: Protective Mechanical VENTilation Strategy in Patients Undergoing CARDiac Surgery (VENT CARD Trial)
Brief Title: Protective Mechanical VENTilation Strategy in Patients Undergoing CARDiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Manager Anesthesia Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-5171
Record Dates: First submitted 2017-09-12; First posted 2017-09-20 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Complications; Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects randomized to the intervention group will receive a comprehensive perioperative mechanical ventilation strategy that includes a bundle of protective settings (use of PEEP, recruitment maneuvers and continuation of mechanical ventilation during CPB).
  Interventions: Other: A comprehensive perioperative mechanical ventilation strategy
- Control Group (No Intervention): Subjects randomized to the control group will receive mechanical ventilation according to the current usual care.

INTERVENTIONS:
Other: A comprehensive perioperative mechanical ventilation strategy — 1) Intervention group.
  * Recruitment maneuvers (doubling the tidal volumes for 10 consecutive breaths) every 30min and after every time mechanical ventilation is stopped for surgical reasons, suctioning occurs or the breathing circuit is disconnected
  * Mechanical ventilation will be continued during CPB (PEEP 5 cm H2O, respiratory rate 8/min, Tidal Volume 6 ml/kg PBW, FiO2 21%
  * Avoidance of lung de-recruitment during patient's transfer (use of PEEP via PEEP valves, endotracheal tube clamps during disconnection from the breathing circuit)
  * Avoidance of disconnection from respiratory circuit during respiratory secretions suctioning (applying closed suction circuits)
  * For the remaining aspects the mechanical ventilation settings will be the same as in the control group.
  Tidal volume 6ml/kg PBW PEEP 5cm H20 FiO2 to target SatO2 of 92-97% Discontinuation of mechanical ventilation during cardiopulmonary bypass
  Arms: Intervention Group

SUMMARY:
Heart surgery is a life-saving intervention for hundreds of thousands of patients each year worldwide. Advances in technology and medical expertise have improved outcomes for these patients over the years. However, despite such advances, approximately 30% of patients develop lung complications (also called "pulmonary complications") after heart surgery, which result in prolonged hospital stay, increased mortality and healthcare costs.

During and immediately after heart surgery, the patient's breathing needs to be artificially controlled by a breathing machine, called "mechanical ventilator". The medical literature has reported that in critically ill patients the use of specific settings on the breathing machine (so called "protective mechanical ventilation") prevents lung complications and significantly decreases mortality. Studies show that such settings could also be beneficial for patients that undergo several types of planned surgery, however data regarding heart surgery patients (the most vulnerable to lung complications) are lacking.The aim of our study is to test whether the use of protective mechanical ventilation settings during and after heart surgery reduces lung complications compared to the current standard of care. The main innovation of this study is the application of a novel protective mechanical ventilation strategy to patients undergoing cardiac surgery, in order to reduce post-operative pulmonary complications.

DETAILED DESCRIPTION:
Postoperative pulmonary complications are frequent after cardiac surgery, affecting approximately 30% of all patients. Such complications result in increased morbidity, mortality and health care utilization. During and immediately after surgery, mechanical ventilation is required to control the patient's breathing. Recent scientific literature showed the striking importance of specific mechanical ventilation settings (which often constituted a bundle of interventions and were generally called "protective mechanical ventilation") in other areas of medicine (i.e., critical care, abdominal surgery, management of organ donors) to prevent the onset or propagation of lung injury as well as multiple organ dysfunction. These protective settings include tidal volume of 6 ml/kg of ideal body weight (as opposed to the traditional tidal volume of 10-12 ml/kg), use of positive end expiratory pressure (PEEP), recruitment maneuvers (temporary periodic application of higher respiratory pressures or volumes on the mechanical ventilator in order to re-open collapsed areas of the lungs) and attention at avoiding lung collapse during patient transfer and suctioning (i.e. maintaining PEEP during transfer and avoiding disconnection from the breathing circuit during suctioning of respiratory secretions). Such interventions could play an even more important role during cardiac surgery, where several insults to the lung take place. These insults result from the inflammatory cascade triggered by cardiopulmonary bypass (CPB), myocardial injury and areas of lung collapse (atelectasis). Indeed, a recent retrospective study showed that the tidal volume utilized during and after cardiac surgery impacts significantly on organ dysfunction, with a tidal volume less than 10 ml/kg of ideal body weight providing better outcomes than larger tidal volumes.

The investigators hypothesize that our proposed bundle of protective mechanical ventilation settings aimed at minimizing lung injury by continuation of mechanical ventilation during cardiopulmonary bypass, recruitment maneuvers, and use of systems that prevent lung collapse during patient transfer and suctioning (i.e. PEEP valves and closed respiratory circuits) will reduce postoperative pulmonary complications compared to the current standard of care, hence significantly improving patients outcomes and reducing health care costs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Scheduled for elective Coronary Artery Bypass Graft, Single valve repair or replacement, or Coronary Artery Bypass Graft plus Single Valve repair or replacement, with the use of Cardiopulmonary Bypass (CPB), aortic clamp and cardioplegia, sternotomy

Exclusion Criteria:

* Pregnancy
* Clinically significant Congenital Heart Disease
* Surgery with planned thoracotomy approach with one lung ventilation
* Body mass index (the weight in kilograms divided by the square of the height in meters) of 40 or higher,
* Receipt of positive pressure mechanical ventilation (invasive and non-invasive) within the 2 weeks preceding surgery (excluding routine treatment for obstructive sleep apnea syndrome)
* Severe chronic respiratory disease, as indicated by any of:
* Baseline FEV1 < 20 ml/kg predicted body weight
* Pre-existing chronic interstitial lung disease with chronic interstitial infiltration on chest X-ray
* Documented chronic CO2 retention (PaCO2 > 50 mm Hg) and/or chronic hypoxaemia (PaO2<55 mmHg on FiO2 = 0.21)
* Chronic restrictive, obstructive, neuromuscular, chest wall or pulmonary vascular disease resulting in severe exercise restriction (e.g., unable to climb stairs or perform household duties), secondary polycythaemia, severe pulmonary hypertension (mean PAP > 40 mmHg), or ventilator dependency
* Requirement for urgent/emergent surgery
* Progressive neuromuscular illness* that will result in prolonged need for mechanical ventilation
* Previous randomization in this trial
* Consent refusal
* Surgeon, anesthesiologist, intensivist refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pulmonary complications | for 7 days post operatively
  Daily chart review and assessment of any pulmonary complications documented

SECONDARY OUTCOMES:
Ventilator free days | Post op day 1-28 days
  number of days without a ventilator
  Number of days without ventilation
Intensive care length of stay | Post op day 1-28 days
  Number of days in the intensive care unit
Hospital length of stay | Post op day 1-28 days
  Number of days in the hospital
Duration of mechanical ventilation | Post op day 1-28 days
  Length of time on a ventilator
Ease of surgical access | Intraoperatively during surgery
  Ability of the surgeon to access the surgical field during cardiopulmonary bypass using a 5 point Likert scale
Barotrauma | in the first 7 days after surgery
  defined as radiological evidence of pneumothorax and/or pneumomediastinum
Surgical complications | From the day of surgery to 48 hours post surgery
  death, myocardial infarction, stroke, acute liver injury, and chest reopening
Acute Kidney Injury | Day of surgery to 28 days
  Incidence of Acute Kidney Injury across the study population
Mortality | Day of surgery to 90-day
  Incidence of mortality across the study population
Home and alive | up to 30 days after surgery
  to evaluate days at home

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Parotto, MD, PhD, Principal Investigator — Toronto General Hospital, UHN
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No